CLINICAL TRIAL: NCT02221830
Title: Postpartum Hemorrhage Prevention in Patients With Preeclampsia (PHP3 Study)
Acronym: PHP3
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-2738; UL1TR001082 (NIH)
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal Saline (standard of care)
  Interventions: Drug: Placebo
- Treatment (Experimental): normal saline + oxytocin
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Our intervention simply replaces the standardly given normal saline with treatment (normal saline + oxytocin)
  Arms: Treatment
Drug: Placebo — This intervention utilizes a Placebo Camparator
  Arms: Placebo

SUMMARY:
Evaluation of the efficacy of postpartum 24 hour oxytocin infusion to reduce blood loss in patients with pre-eclampsia (PE)

DETAILED DESCRIPTION:
The overall goal of this study is to evaluate the efficacy of postpartum 24 hour oxytocin infusion as a prevention-oriented strategy to reduce blood loss in patients with pre-eclampsia (PE) in a blinded, placebo controlled, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. vaginal or cesarean delivery at a gestational age greater than or equal to 20 weeks gestational age;
2. diagnosis of preeclampsia (PE defined using standard definitions based on the ACOG bulletin and the NIH Working Group on High Blood Pressure in Pregnancy (i.e., a systolic blood pressure greater than 140 mm Hg or a diastolic blood pressure greater than 90 mm Hg on at least 2 occasions at least 6 hours apart after 20 weeks gestation and proteinuria of > 300mg per 24 hour period or > 1+ on dipstick).
3. patients treated with magnesium sulfate for 24 hours post partum at 2g/hr (standard of care when deemed appropriate by clinician for seizure prophylaxis)

Exclusion Criteria:

1. abnormal placentation (previa, accreta, etc)
2. antenatal hemorrhage
3. contraindication to oxytocin

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02; Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of Postpartum hematocrit | 24 hours postpartum
  Postpartum hematocrit (collected 24 hours after delivery unless patient receives blood transfusion, then pre-transfusion hematocrit will be used)

SECONDARY OUTCOMES:
Primary postpartum hemorrhage | Before discharge from hospital
  Considered to be >500ml with vaginal deliveries,or, >1000ml with cesarean sections.
Estimated blood loss at delivery | Before discharge from hospital
  Estimated blood loss at delivery
Postpartum blood loss | 24 hours postpartum
  Postpartum blood loss: 24hrs postpartum, as measured by pad counts and weights.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Hermesch, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Clinical and Translational Research Center, Aurora, Colorado, United States